CLINICAL TRIAL: NCT04095481
Title: Obalon Navigation/Touch System Post-Approval Study
Acronym: NTS PAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Obalon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-7410-0007
Record Dates: First submitted 2019-08-26; First posted 2019-09-19 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Obalon NTS: Patients who commercially purchased the NTS Compatible Obalon Balloon System
  Interventions: Device: Obalon Navigation/Touch System

INTERVENTIONS:
Device: Obalon Navigation/Touch System — The NTS Compatible Obalon Balloon System does NOT require the use of radiographic verification prior to the inflation of the intragastric balloon

SUMMARY:
Post-approval study for the Obalon Navigation/Touch System (NTS)

DETAILED DESCRIPTION:
The Obalon NTS PAS is a prospective, observational, open-label and multi-center study with an objective to collect continued safety and performance of the Obalon NTS in a commercial setting and confirm results observed in the supplemental PMA IDE study.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 22 years and older
2. Starting or current therapy BMI of 30.0-40.0 kg/m2
3. Commercially purchased the Obalon Balloon Device

Exclusion Criteria:

1. Known history of structural or functional disorders of the esophagus that may impede passage of the device through the gastrointestinal tract or increase risk of esophageal damage during an endoscopic removal procedure, including, Barrett's esophagus, esophagitis, dysphagia, achalasia, stricture/stenosis, esophageal varices, esophageal diverticula, esophageal perforation or any other disorder of the esophagus.
2. Known history of structural or functional disorder of the esophagus, including any swallowing disorder, esophageal chest pain disorders, or drug refractory esophageal reflux symptoms.
3. Known history of structural or functional disorders of the stomach including, gastroparesis, gastric ulcer, chronic gastritis, gastric varices, hiatal hernia (> 2 cm), cancer or any other disorder of the stomach.
4. Active implantable devices, such as a pacemaker of defibrillator, or with metal implants in the thoracic region.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 22 years and older with a starting therapy BMI of 30.0-40.0 kg/m2 and who commercially purchased the Obalon Balloon device.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Esophageal Inflation | Up to 20 Weeks
  Percentage of esophageal Inflation during the balloon administrations using the Obalon NTS.
System Success | Up to 20 Weeks
  Percentage of appropriate inflation in the stomach with the use of NTS only (without radiography) or correctly determining failed balloon transit (device in the esophagus) as confirmed by endoscopic removal

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ultimate Bariatrics - Flower Mound, Flower Mound, Texas
  - Ultimate Bariatrics - Fort Worth, Fort Worth, Texas